CLINICAL TRIAL: NCT03180515
Title: Neural and Kinematic Features of Freezing of Gait for Adaptive Neurostimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Helen M. Bronte-Stewart, John E. Cahill Family Profressor, Professor of Neurology and, by courtesy, Neurosurgery at the Stanford University Medical Center, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1R21NS096398 (NIH)
Record Dates: First submitted 2017-06-06; First posted 2017-06-08 (Actual); Results first posted 2019-11-04 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Activa PC+S Neurostimulator (Experimental): All patients will complete motor testing on both continuous DBS and adaptive DBS during a study visit. The UPDRS rater and the patient will be blind to which type of stimulation they are on.
  Interventions: Device: Activa PC+S Neurostimulator

INTERVENTIONS:
Device: Activa PC+S Neurostimulator — Activa PC+S Neurostimulator is approved for both aDBS and cDBS paradigms.
  Other Names: adaptive deep brain stimulation (aDBS); continuous deep brain stimulation (cDBS)

SUMMARY:
Continuous deep brain stimulation (cDBS) is an established therapy for the major motor signs in Parkinson's disease, however some patients find that it does not adequately treat their freezing of gait (FOG). Currently, cDBS is limited to "open-loop" stimulation,without real-time adjustment to the patient's state of activity, fluctuations and types of motor symptoms, medication dosages, or neural markers of the disease. The purpose of this study is to determine if an adaptive DBS system,responding to patient specific, clinically relevant neural or kinematic feedback related to FOG, is more effective than continuous DBS on the motor Unified Parkinson's Disease Rating Scale (UPDRS III) and gait measures of PD.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of idiopathic Parkinson's disease, with bilateral symptoms at Hoehn and Yahr Stage greater than or equal to II.
2. Documented improvement in motor signs on versus off dopaminergic medication, with a change in the Unified Parkinson's Disease Rating Scale motor (UPDRS III) score of >= 30% off to on medication.
3. The presence of complications of medication such as wearing off signs,fluctuating responses and/or dyskinesias, and/or medication refractory tremor,and/or impairment in the quality of life on or off medication due to these factors.
4. Subjects should be on stable doses of medications, which should remain unchanged until the DBS system is activated. After the DBS system is optimized(during which time the overall medication dose may be reduced to avoid discomfort and complications such as dyskinesias) the medication dose should remain unchanged, if possible, for the duration of the study.
5. Treatment with carbidopa/levodopa, and with a dopamine agonist at the maximal tolerated doses as determined by a movement disorders neurologist.
6. Ability and willingness to return for study visits, at the initial programming and after three, six and twelve months of DBS.
7. Age > 18
8. Has a history of and/or displays freezing of gait

Exclusion Criteria:

1. Subjects with significant cognitive impairment and/or dementia as determined bya standardized neuropsychological battery.
2. Subjects with clinically active depression, defined according to the Diagnostic and Statistical manual of Mental Disorders, Fourth Edition (DSM-IV) criteria and as scored on a validated depression assessment scale.
3. Subjects with very advanced Parkinson's disease, Hoehn and Yahr stage 5 on medication (non-ambulatory).
4. Age > 80.
5. Subjects with an implanted electronic device such as a neurostimulator, cardiac pacemaker/defibrillator or medication pump.
6. Subjects, who are pregnant, are capable of becoming pregnant, or who are breast feeding.
7. Patients with cortical atrophy out of proportion to age or focal brain lesions that could indicate a non-idiopathic movement disorder as determined by MRI
8. Subjects having a major comorbidity increasing the risk of surgery (prior stroke,severe hypertension, severe diabetes, or need for chronic anti-coagulation other than aspirin).
9. Subjects having any prior intracranial surgery.
10. Subjects with a history of seizures.
11. Subjects, who are immunocompromised.
12. Subjects with an active infection.
13. Subjects, who require diathermy, electroconvulsive therapy (ECT), or transcranial magnetic stimulation (TMS) to treat a chronic condition.
14. Subjects, who have an inability to comply with study follow-up visits or study protocol.
15. Subjects, who are unable to understand or sign the informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen Bronte-Stewart, MS, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Movement Disorders, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Activa PC+S Neurostimulator: For Aim 1, all participants participated in the same "state" - off dopaminergic medication and off deep brain stimulation (DBS), so that we could characterize the two groups (freezers and non-freezers, respectively people who experience freezing of gait and those who do not) at baseline.
  For Aim 2, all participants underwent randomized presentations of OFF, 60 Hz DBS and 140 Hz DBS while completing several walking tasks. (So all participants had walking trials off stimulatoin, all had walking trials at 60 Hz DBS, all had walking trials at 140 Hz DBS).
  For Aim 3, due to technological limitations and resources, only one subject completed the stepping in place task while on continuous DBS (cDBS), and completed the stepping in place task again while on adaptive DBS (aDBS).
  For Aim 3, Aim 1 Arms: Freezers vs. non-freezers Aim 2 Arms: OFF vs. 60 Hz DBS vs. 140 Hz DBS Aim 3 Arms: OFF vs. cDBS vs. aDBS
Period: Aim 1
Arm/Group | Activa PC+S Neurostimulator
Started | 12
Completed | 12
Not Completed | 0
Period: Aim 2
Arm/Group | Activa PC+S Neurostimulator
Started | 12
Completed | 12
Not Completed | 0
Period: Aim 3
Arm/Group | Activa PC+S Neurostimulator
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Activa PC+S Neurostimulator: All patients
Arm/Group | Activa PC+S Neurostimulator
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.27 (7.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Unified Parkinson's Disease Rating Scale III Score (OFF) [Mean (Standard Deviation); unit: units on a scale] — The Unified Parkinson's Disease Rating Scale or UPDRS Part III is the motor examination of the standard clinical rating scale used to gauge the course of Parkinson's disease in patients. Total score is reported as the sum of the subscores, and higher values indicate greater disease severity. The range for the total score of the UPDRS III Motor Examination is between 0-108.
  units on a scale | 34.8 (14.8)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] Related to aDBS
Description: Safety, tolerability and feasibility of aDBS
Time Frame: 30 min - 2 hours
Population: Due to limitations in technology and resources we were only able to test a single participant during the stepping in place task while on continuous DBS and while on adaptive DBS.
Measure: Number; unit: Number of Treatment Emergent AEs
Groups:
- (OFF) Activa PC+S Neurostimulator: OFF stimulation
- (cDBS) Activa PC+S Neurostimulator: Continuous or open-loop DBS
- (aDBS) Activa PC+S Neurostimulator: Adaptive DBS
Arm/Group | (OFF) Activa PC+S Neurostimulator | (cDBS) Activa PC+S Neurostimulator | (aDBS) Activa PC+S Neurostimulator
Number analyzed (Participants) | 1 | 1 | 1
Number of Treatment Emergent AEs | 0 | 0 | 0

2. Secondary Outcome: Aim 1: Alpha Power
Description: Subthalamic nucleus (STN) local field potentials (LFP) recordings demonstrate oscillatory neuronal activity in both the alpha (8-12 Hz) and beta (13-30 Hz) bands in the resting state in PD. Spectrograms were generated using a short-time Fourier transform, with a 1 second Hanning window and a 0.5 second overlap, creating a frequency resolution of 1 Hz. Power spectral densities were calculated using the Welch method with the same window and overlap parameters. Power was summed in the beta and alpha bands. This power can be representative of the magnitude of oscillatory activity in this frequency band occurring in this brain region.
Time Frame: 30 minutes
Population: Subjects were classified as a Freezer or Non-Freezer by the clinical history of a subject's symptoms and/or if the subject displayed freezing behavior pre-operatively or during the tasks.
Measure: Mean (Standard Deviation); unit: arbitrary units (power)
Groups:
- Freezers: PD subjects with Freezing of Gait
- Non-Freezers: PD subjects without Freezing of Gait
Arm/Group | Freezers | Non-Freezers
Number analyzed (Participants) | 8 | 4
arbitrary units (power)
  Stepping in Place Task | 0.845 (0.543) | 1.051 (0.511)
  Forward Walking | 1.710 (1.280) | 2.753 (3.261)
  Turning and Barrier Course | 1.393 (0.901) | 1.890 (1.351)

3. Secondary Outcome: Aim 1: Beta Power
Description: as for outcome 2
Time Frame: 30 minutes
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: arbitrary units (power)
Arm/Group | Freezers | Non-Freezers
Number analyzed (Participants) | 8 | 4
arbitrary units (power)
  Stepping in Place Task | 4.085 (2.077) | 11.258 (8.493)
  Forward Walking | 9.143 (6.835) | 8.400 (5.529)
  Turning and Barrier Course | 7.321 (4.429) | 6.993 (0.207)

4. Secondary Outcome: Aim 1: Alpha Sample Entropy
Description: The predictability of the local field potentials (band-pass filtered between 8-12 Hz for alpha) was analyzed using Sample Entropy (SampEn), a nonlinear measure suitable for physiological time series. SampEn may be a more consistent measure and more suitable to shorter time series data than approximate entropy, partially due to the elimination of counting self matches. SampEn is calculated as the negative logarithm of the estimated conditional probability that if consecutive subseries of length m are similar according to some preset tolerance r, the consecutive subseries of length m+1 will be similar too. Here the length of the vector pairs, m, denotes the embedding dimension.
Time Frame: 30 minutes
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Freezers | Non-Freezers
Number analyzed (Participants) | 8 | 4
arbitrary units
  Stepping in Place Task | 0.251 (0.002) | 0.253 (0.004)
  Forward Walking | 0.248 (0.007) | 0.247 (0.007)
  Turning and Barrier Course | 0.253 (0.003) | 0.250 (0.004)

5. Secondary Outcome: Aim 1: Beta Sample Entropy
Description: The predictability of the local field potentials (band-pass filtered between 15-30 Hz for beta) was analyzed using Sample Entropy (SampEn), a nonlinear measure suitable for physiological time series. SampEn may be a more consistent measure and more suitable to shorter time series data than approximate entropy, partially due to the elimination of counting self matches. SampEn is calculated as the negative logarithm of the estimated conditional probability that if consecutive subseries of length m are similar according to some preset tolerance r, the consecutive subseries of length m+1 will be similar too. Here the length of the vector pairs, m, denotes the embedding dimension.
Time Frame: 30 minutes
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Freezers | Non-Freezers
Number analyzed (Participants) | 8 | 4
arbitrary units
  Stepping in Place Task | 0.407 (0.031) | 0.337 (0.062)
  Forward Walking | 0.380 (0.050) | 0.376 (0.053)
  Turning and Barrier Course | 0.377 (0.050) | 0.376 (0.052)

6. Secondary Outcome: Aim 2: Asymmetry
Description: Asymmetry during both forward walking and stepping in place was calculated using periods of walking or stepping when the subject was not freezing. According to previous studies, asymmetry is defined as: 100*(absolute value of the natural log of the shorter average swing time over the longer average swing time) or mathematically: 100*| ln (SSWT/LSWT) |
  where SSWT = shorter mean swing time LSWT = longer mean swing time
Time Frame: 30 minutes
Population: 12 participants total: the 8 freezers are the same participants across stimulation conditions; the 4 non-freezers are the same participants across stimulation conditions. Subjects were classified Freezer/Non-Freezer by the clinical history of a subject's symptoms and/or if the subject displayed freezing behavior pre-operatively or during the tasks.
Measure: Mean (Standard Deviation); unit: asymmetry (%)
Groups:
- Freezers (OFF Stim): PD subjects with Freezing of Gait OFF Stimulation
- Freezers (60 Hz Stim): PD subjects with Freezing of Gait on 60 Hz Stimulation
- Freezers (140 Hz Stim): PD subjects with Freezing of Gait on 140 Hz Stimulation
- Non-Freezers (OFF Stim): PD subjects without Freezing of Gait OFF Stimulation
- Non-Freezers (60 Hz Stim): PD subjects without Freezing of Gait on 60 Hz Stimulation
- Non-Freezers (140 Hz Stim): PD subjects without Freezing of Gait on 140 Hz Stimulation
Arm/Group | Freezers (OFF Stim) | Freezers (60 Hz Stim) | Freezers (140 Hz Stim) | Non-Freezers (OFF Stim) | Non-Freezers (60 Hz Stim) | Non-Freezers (140 Hz Stim)
Number analyzed (Participants) | 8 | 8 | 8 | 4 | 4 | 4
asymmetry (%)
  Stepping in Place Task | 26.74 (23.44) | 27.1 (21.42) | 15.99 (12.12) | 9.54 (6.87) | 7.86 (7.10) | 7.25 (9.03)
  Forward Walking | 6.11 (4.11) | 5.01 (2.97) | 4.52 (3.39) | 3.32 (1.88) | 2.41 (2.50) | 4.50 (2.23)

7. Secondary Outcome: Aim 2: Arrhythmicity
Description: Arrhythmicity during both forward walking and stepping in place was calculated using periods of walking or stepping when the subject was not freezing. According to previous studies, arrhythmicity is defined as the mean stride time coefficient of variation of both legs, and a greater stride time CV implies less rhythmic gait or stepping. Higher arrhythmicity corresponds to more arrhythmic, or more impaired, gait.
Time Frame: 30 minutes
Population: 12 participants total: the 8 freezers are the same participants across stimulation conditions; the 4 non-freezers are the same participants across stimulation conditions.
Measure: Mean (Standard Deviation); unit: arrythmicity (CV%)
Arm/Group | Freezers (OFF Stim) | Freezers (60 Hz Stim) | Freezers (140 Hz Stim) | Non-Freezers (OFF Stim) | Non-Freezers (60 Hz Stim) | Non-Freezers (140 Hz Stim)
Number analyzed (Participants) | 8 | 8 | 8 | 4 | 4 | 4
arrythmicity (CV%)
  Stepping in Place Task | 54.04 (50.46) | 27.49 (33.23) | 29.34 (56.18) | 4.01 (0.81) | 4.10 (1.40) | 4.00 (0.73)
  Forward Walking | 6.76 (3.29) | 5.18 (2.25) | 6.41 (2.68) | 5.98 (4.37) | 4.96 (1.35) | 4.94 (1.38)

8. Secondary Outcome: Aim 2: Stride Time
Description: Kinematic Features associated with Freezing of Gait
Time Frame: 30 minutes
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Freezers (OFF Stim) | Freezers (60 Hz Stim) | Freezers (140 Hz Stim) | Non-Freezers (OFF Stim) | Non-Freezers (60 Hz Stim) | Non-Freezers (140 Hz Stim)
Number analyzed (Participants) | 8 | 8 | 8 | 4 | 4 | 4
seconds
  Stepping in Place Task | 1.71 (0.68) | 1.44 (0.53) | 1.21 (0.44) | 1.07 (0.15) | 1.05 (0.14) | 1.06 (0.17)
  Forward Walking | 1.14 (0.19) | 1.11 (0.15) | 1.10 (0.14) | 1.16 (0.06) | 1.15 (0.07) | 1.18 (0.10)

9. Secondary Outcome: Aim 2: Percent Time Freezing
Description: Freezing of gait episodes during stepping in place were identified using a validated computerized algorithm, and during forward walking by a blinded rater. The percent time freezing was calculated by dividing the time spent freezing by the total time to complete the task then multiplying by 100 to get a percent. If no freezing was observed, then the percent time freezing reported was 0.0%.
Time Frame: 30 minutes
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: % time freezing
Arm/Group | Freezers (OFF Stim) | Freezers (60 Hz Stim) | Freezers (140 Hz Stim) | Non-Freezers (OFF Stim) | Non-Freezers (60 Hz Stim) | Non-Freezers (140 Hz Stim)
Number analyzed (Participants) | 8 | 8 | 8 | 4 | 4 | 4
% time freezing
  Stepping in Place Task | 29.37 (38.27) | 11.01 (29.57) | 18.13 (34.58) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  Forward Walking | 0.17 (0.48) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)

10. Secondary Outcome: Percent Time Freezing
Description: Freezing of gait episodes during stepping in place were identified using a validated computerized algorithm. The percent time freezing was calculated by dividing the time spent freezing by the total time to complete the task then multiplying by 100 to get a percent. If no freezing was observed, then the percent time freezing reported was 0.0%. The percent time spent freezing was compared while the participant was doing the stepping in place task on continuous deep brain stimulation (cDBS) and while the participant was doing the stepping in place task on adaptive deep brain stimulation (aDBS).
Time Frame: 30 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % time freezing
Arm/Group | (OFF) Activa PC+S Neurostimulator | (cDBS) Activa PC+S Neurostimulator | (aDBS) Activa PC+S Neurostimulator
Number analyzed (Participants) | 1 | 1 | 1
% time freezing | 44 (0) | 2 (0) | 0 (0)

ADVERSE EVENTS:
Time Frame: 2 days - throughout the entirety of the research visit
Description: No AE's reported. We used an adverse events questionnaire to assess whether patients felt any of the following: pins and needles, tightness in arm or face, light headedness, nausea, speech problems, confusion/cognitive changes, unwanted mood changes, balance problems, other symtpoms/notes.
Groups:
- Activa PC+S Neurostimulator Aim 1: Aim 1 Arms: Freezers vs. non-freezers All participants participated in Aim 1
- Activa PC +S Neurostimulator Aim 2: Aim 2 Arms: OFF vs. 60 Hz DBS vs. 140 Hz DBS
  All participants participated in Aim 2.
  Within participant, adverse effects were assessed between OFF DBS, 60 Hz DBS and 140 Hz DBS.
- Activa PC +S Neurostimulator Aim 3: Aim 3 Arms: OFF vs. cDBS vs. aDBS
  Due to limitations in technology and resources, only one participant participated in Aim 3.
  Within participant, adverse effects were assessed between OFF DBS, cDBS, and aDBS.
Arm/Group | Activa PC+S Neurostimulator Aim 1 | Activa PC +S Neurostimulator Aim 2 | Activa PC +S Neurostimulator Aim 3
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/1
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-09-04): https://cdn.clinicaltrials.gov/large-docs/15/NCT03180515/SAP_000.pdf
  • Study Protocol (2018-11-20): https://cdn.clinicaltrials.gov/large-docs/15/NCT03180515/Prot_001.pdf